CLINICAL TRIAL: NCT01009047
Title: A Randomized, Multicenter, Double-Blind, Active-Controlled, Flexible-Dose, Parallel-Group Study of the Efficacy and Safety of Extended Release Paliperidone for the Treatment of Symptoms of Schizophrenia in Adolescent Subjects, 12 to 17 Years of Age
Brief Title: An Efficacy and Safety Study of Extended-Release (ER) Paliperidone in Adolescent Participants With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR016675; R076477PSZ3003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2013-06-21 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone; Aripiprazole
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paliperidone extended-release (ER) (Experimental): Paliperidone ER will be administered as oral capsule at a dose of 6 milligram (mg) for 1 week and then will be administered at a dose of either 3, 6 or 9 mg up to Week 26, once daily in the morning.
  Interventions: Drug: Paliperidone extended release (ER)
- Aripiprazole (Active Comparator): Aripiprazole will be administered as oral capsule at a dose of 2 mg on Days 1 and 2, 5 mg on Days 3 and 4, 10 mg Days 5, 6 and 7; and then will be administered as a dose of either 5 or 10 or 15 mg up to Week 26, once daily in the morning.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Paliperidone extended release (ER) — Paliperidone ER will be administered as oral capsule at a dose of 6 mg for 1 week and then will be administered at a dose of either 3, 6 or 9 mg up to Week 26, once daily in the morning.
  Arms: Paliperidone extended-release (ER)
Drug: Aripiprazole — Aripiprazole will be administered as oral capsule at a dose of 2 mg on Days 1 and 2, 5 mg on Days 3 and 4, 10 mg Days 5, 6 and 7; and then will be administered as a dose of either 5 or 10 or 15 mg up to Week 26, once daily in the morning.
  Arms: Aripiprazole

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of extended-release (ER) paliperidone compared to aripiprazole (atypical antipsychotic) in symptomatic (having symptoms) adolescent participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations [imagining things], and withdrawal into the self) .

DETAILED DESCRIPTION:
This is a multi-center (conducted in more than 1 center), double-blind (neither physician nor participant knows the name of the assigned drug), randomized (study drug is assigned by chance), active-controlled (paliperidone ER is compared to aripiprazole), parallel-group (a medical research study comparing the response in 2 or more groups of participants receiving different treatments), flexible-dose (the physician has the freedom to give different doses to the participant depending on how they respond to treatment) study designed to determine the efficacy and safety of paliperidone ER in symptomatic adolescents (12 to 17 years of age) with schizophrenia. The total duration of the study will be approximately 29 weeks. The study consists of 3 phases: a Screening phase up to 3 weeks (with a possible overlapping washout period), a Double-blind acute phase of 8 weeks, and a Double-blind maintenance phase of 18 weeks. Participants will be randomly assigned to 1 of the 2 treatment groups (paliperidone ER or aripiprazole flexible oral doses). Dosage will be adjusted at the scheduled visits. Efficacy of the participants will primarily be evaluated through Positive and Negative Syndromes Scale (PANSS). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must currently meet the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria for schizophrenia and have experienced symptoms of the illness for at least 1 year, and they should have had at least treatment with 1 antipsychotic before participation in this study
* Participants having a Positive and Negative Syndromes Scale (PANSS) score between 60 and 120 inclusive at Screening
* Female participants must be incapable of pregnancy, or if heterosexually active and capable of pregnancy, have been using an acceptable method of contraception for at least 1 month before study entry and agree to continue use contraception methods for the duration of the study, or if sexually abstinent (not having sexual intercourse) and capable of pregnancy, must agree to continue abstinence or to use an acceptable method of birth control
* Participants must not be a danger to themselves or others, and must have family support available to be maintained as out-patients
* Participants with a weight of equal to or greater than 29 kilogram

Exclusion Criteria:

* Participants with mild (not serious), moderate (medium level of seriousness), or severe (very serious, life threatening) mental retardation
* Participants with a known or suspected history of substance dependence (including alcohol, but excluding nicotine or caffeine) as per the DSM-IV criteria in the 3 months before Screening
* Participants with a history of certain neurological (pertaining to the nervous system) disorders or insulin-dependent diabetes mellitus (disorder in which there is decreased insulin in the body or the body's insulin is not effective, resulting in high blood sugar, increased thirst and urine, and many other side effects)
* Participants who have received a depot injectable antipsychotic within 2 treatment cycles before the Screening visit
* Participants who have received clozapine in 2 months before the Baseline visit (Day 1 of Week 1)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 228 (Actual)
Dates: Start 2009-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (41):
- United States (6):
  - Dothan, Alabama
  - Santa Ana, California
  - Atlanta, Georgia
  - Smyrna, Georgia
  - Lake Charles, Louisiana
  - Shreveport, Louisiana
- India (5):
  - Jaipur
  - Kanpur Uttarpradeh
  - Lucknow Gpo
  - Mangalore
  - Varanasi
- Bucharest, Romania
- Russia (13):
  - Chelyabinsk
  - Ekaterinburg Na
  - Krasnodar
  - Moscow
  - Moscow Russia
  - Nizhny Novgorod
  - Novosibirsk
  - Saint Petersburg
  - Samara
  - Saratov
  - Smolensk Region N/A
  - Tomsk Na
  - Yaroslavl
- Bratislava, Slovakia
- Spain (7):
  - Badajoz
  - Esplugues de Llobregat
  - Madrid
  - Paterna
  - Sabadell
  - Seville
  - Valladolid
- Ukraine (8):
  - Donetsk
  - Hlevakha
  - Ivano-Frankivsk
  - Kharkiv
  - Kherson
  - Kiev
  - Poltava
  - Simferopol

REFERENCES:
- [Derived] Savitz AJ, Lane R, Nuamah I, Gopal S, Hough D. Efficacy and safety of paliperidone extended release in adolescents with schizophrenia: a randomized, double-blind study. J Am Acad Child Adolesc Psychiatry. 2015 Feb;54(2):126-137.e1. doi: 10.1016/j.jaac.2014.11.009. Epub 2014 Nov 25. PMID 25617253

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone Extended Release (ER): Paliperidone ER administered as oral capsule at a dose of 6 milligram (mg) for 1 week and then administered at a dose of either 3, 6 or 9 mg up to Week 26, once daily in the morning.
- Aripiprazole: Aripiprazole administered as oral capsule at a dose of 2 mg on Days 1 and 2, 5 mg on Days 3 and 4; 10 mg on Days 5, 6 and 7; and then administered as a dose of either 5 or 10 or 15 mg up to Week 26, once daily in the morning.
Period: Overall Study
Arm/Group | Paliperidone Extended Release (ER) | Aripiprazole
Started | 113 | 115
Completed | 85 | 89
Not Completed | 28 | 26
Not completed — Adverse Event | 5 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Lack of Efficacy | 4 | 11
Not completed — Withdrawal by consent | 16 | 11
Not completed — Other | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Paliperidone Extended Release (ER): Paliperidone ER administered as oral capsule at a dose of 6 mg for 1 week and then administered at a dose of either 3, 6 or 9 mg up to Week 26, once daily in the morning.
- Total: Total of all reporting groups
Arm/Group | Paliperidone Extended Release (ER) | Aripiprazole | Total
Number analyzed (Participants) | 112 | 114 | 226
Age Continuous [Mean (Standard Deviation); unit: Years] — Number of participants analyzed for this Baseline characteristic is intent to treat (ITT) population which included all randomly assigned participants who received at least 1 dose of double-blind study drug, had both a Baseline measurement and at least 1 Post-Baseline measurement in the double-blind phase. Last observation carried forward (LOCF) method was used.
  Years | 15.3 (1.46) | 15.4 (1.45) | 15.3 (1.46)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of participants analyzed for this Baseline characteristic is intent to treat (ITT) population which included all randomly assigned participants who received at least 1 dose of double-blind study drug, had both a Baseline measurement and at least 1 Post-Baseline measurement in the double-blind phase. Last observation carried forward (LOCF) method was used.
  Participants
    Female | 39 | 38 | 77
    Male | 73 | 76 | 149

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score at Day 56
Description: The PANSS is a 30-item scale with each item rated on a scale of 1 (absent) to 7 (extreme psychopathology), designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening.
Time Frame: Baseline and Day 56
Population: The intent-to-treat (ITT) population included all randomly assigned participants who received at least 1 dose of double-blind study drug, had both a Baseline measurement and at least 1 Post-Baseline measurement in the double-blind phase. Last observation carried forward (LOCF) method was used.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER) | Aripiprazole
Number analyzed (Participants) | 112 | 114
Units on a scale
  Baseline | 89.6 (12.22) | 92.0 (12.09)
  Change at Day 56 | -19.3 (13.80) | -19.8 (14.56)
Statistical Analysis 1: Comparison: Paliperidone Extended Release (ER) vs Aripiprazole; Test type: Superiority or Other; p = 0.935, ANCOVA — Analysis of covariance (ANCOVA) model with treatment (paliperidone ER, aripiprazole) and country as factors, and baseline value as a covariate was used; Least-squares (LS) mean difference = 0.1, 95% CI 2-sided [-3.46 to 3.76], Standard Error of Mean 1.83

2. Secondary Outcome: Change From Baseline in PANSS Total Score at Day 182
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening.
Time Frame: Baseline and Day 182
Population: The ITT population included all randomly assigned participants who received at least 1 dose of double-blind study drug, had both a Baseline measurement and at least 1 Post-Baseline measurement in the double-blind phase. Last observation carried forward (LOCF) method was used.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER) | Aripiprazole
Number analyzed (Participants) | 112 | 114
Units on a scale
  Baseline | 89.6 (12.22) | 92.0 (12.09)
  Change at Day 182 | -25.6 (16.88) | -26.8 (18.82)
Statistical Analysis 1: Comparison: Paliperidone Extended Release (ER) vs Aripiprazole; Test type: Superiority or Other; p = 0.877, ANCOVA — Analysis of covariance (ANCOVA) model with treatment groups (paliperidone ER, aripiprazole) and country as factors, and baseline value as a covariate was used; LS mean difference = -0.3, 95% CI 2-sided [-4.68 to 4.00], Standard Error of Mean 2.20

3. Secondary Outcome: Change From Baseline in Marder Factor Negative Symptoms Score at Day 56 and 182
Description: The PANSS negative subscale based on marder factor assesses 7 negative-symptoms of schizophrenia. Negative symptoms represent a diminution or loss of normal functions. The symptoms are rated on a 7-point scale, with a range of 7 (absent) to 49 (extreme psychopathology).
Time Frame: Baseline, Day 56 and Day 182
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER) | Aripiprazole
Number analyzed (Participants) | 112 | 114
Units on a scale
  Baseline | 23.2 (4.92) | 23.3 (4.54)
  Change at Day 56 | -4.3 (4.56) | -4.7 (4.61)
  Change at Day 182 | -6.0 (5.51) | -6.2 (5.84)
Statistical Analysis 1: Comparison: Paliperidone Extended Release (ER) vs Aripiprazole; Test type: Superiority or Other; p = 0.341, ANCOVA — Day 56: Analysis of covariance (ANCOVA) model with treatment (paliperidone ER, aripiprazole) and country as factors, and baseline value as a covariate was used; LS mean difference = 0.5, 95% CI 2-sided [-0.55 to 1.59], Standard Error of Mean 0.54
Statistical Analysis 2: Comparison: Paliperidone Extended Release (ER) vs Aripiprazole; Test type: Superiority or Other; p = 0.723, ANCOVA — Day 182: Analysis of covariance (ANCOVA) model with treatment (paliperidone ER, aripiprazole) and country as factors, and baseline value as a covariate was used; LS mean difference = 0.2, 95% CI 2-sided [-1.06 to 1.53], Standard Error of Mean 0.66

4. Secondary Outcome: Change From Baseline in Other Marder Factors Scores at Day 56 and 182
Description: The subscales based on marder factors are: positive symptoms, disorganised thoughts factor, uncontrolled hostility/excitement factor, and anxiety/depression factor. The symptoms are rated on a 7-point scale, with a range of 8 to 56 for positive symptoms, 7 to 49 for disorganized thoughts and 4 to 28 for Uncontrolled hostility/excitement and anxiety/depression. Higher score indicate worsening.
Time Frame: Baseline, Day 56 and 182
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER) | Aripiprazole
Number analyzed (Participants) | 112 | 114
Units on a scale
  Baseline: Positive symptoms | 24.6 (4.08) | 24.9 (4.32)
  Change at Day 56: Positive symptoms | -6.1 (4.96) | -5.6 (4.83)
  Change at Day 182: Positive symptoms | -7.8 (5.82) | -7.8 (6.03)
  Baseline: Negative symptoms | 23.2 (4.92) | 23.3 (4.54)
  Change at Day 56: Negative symptoms | -4.3 (4.56) | -4.7 (4.61)
  Change at Day 182: Negative symptoms | -6.0 (5.51) | -6.2 (5.84)
  Baseline: Disorganized thoughts | 21.4 (4.40) | 22.1 (3.86)
  Change at Day 56: Disorganized thoughts | -4.0 (3.34) | -4.1 (3.40)
  Change at Day 182: Disorganized thoughts | -5.5 (4.18) | -5.7 (4.46)
  Baseline: Uncontrolled hostility | 10.7 (3.19) | 11.7 (3.48)
  Change at Day 56: Uncontrolled hostility | -2.5 (2.67) | -2.9 (3.05)
  Change at Day 182: Uncontrolled hostility | -3.2 (3.11) | -3.8 (3.97)
  Baseline: Anxiety/depression | 9.7 (3.17) | 10.0 (3.26)
  Change at Day 56: Anxiety/depression | -2.4 (3.08) | -2.6 (2.81)
  Change at Day 182: Anxiety/depression | -3.0 (3.29) | -3.2 (3.17)
Statistical Analysis 1: Comparison: Paliperidone Extended Release (ER) vs Aripiprazole; Test type: Superiority or Other; p = 0.351, ANCOVA — Change at Day 56: Positive Symptoms - ANCOVA model with treatment groups (paliperidone ER, aripiprazole) and country as factors, and baseline value as a covariate
Statistical Analysis 2: Comparison: Paliperidone Extended Release (ER) vs Aripiprazole; Test type: Superiority or Other; p = 0.691, ANCOVA — Change at Day 182:Positive Symptoms - ANCOVA model with treatment groups (paliperidone ER, aripiprazole) and country as factors, and baseline value as a covariate was used
Statistical Analysis 3: Comparison: Paliperidone Extended Release (ER) vs Aripiprazole; Test type: Superiority or Other; p = 0.965, ANCOVA — Change at Day 56: Disorganized thoughts - ANCOVA model with treatment groups (paliperidone ER, aripiprazole) and country as factors, and baseline value as a covariate was used
Statistical Analysis 4: Comparison: Paliperidone Extended Release (ER) vs Aripiprazole; Test type: Superiority or Other; p = 0.766, ANCOVA — Change at Day 182: Disorganized thoughts - ANCOVA model with treatment groups (paliperidone ER, aripiprazole) and country as factors, and baseline value as a covariate was used
Statistical Analysis 5: Comparison: Paliperidone Extended Release (ER) vs Aripiprazole; Test type: Superiority or Other; p = 0.984, ANCOVA — Change at Day 56: Uncontrolled hostility/ excitement - ANCOVA model with treatment groups (paliperidone ER, aripiprazole) and country as factors, and baseline value as a covariate was used
Statistical Analysis 6: Comparison: Paliperidone Extended Release (ER) vs Aripiprazole; Test type: Superiority or Other; p = 0.985, ANCOVA — Change at Day 182: Uncontrolled Hositility/ Excitement - ANCOVA model with treatment groups (paliperidone ER, aripiprazole) and country as factors, and baseline value as a covariate was used
Statistical Analysis 7: Comparison: Paliperidone Extended Release (ER) vs Aripiprazole; Test type: Superiority or Other; p = 0.803, ANCOVA — Change at Day 56: Anxiety/ depression - ANCOVA model with treatment groups (paliperidone ER, aripiprazole) and country as factors, and baseline value as a covariate
Statistical Analysis 8: Comparison: Paliperidone Extended Release (ER) vs Aripiprazole; Test type: Superiority or Other; p = 0.745, ANCOVA — Change at Day 182: Anxiety/ depression - ANCOVA model with treatment groups (paliperidone ER, aripiprazole) and country as factors, and baseline value as a covariate

5. Secondary Outcome: Change From Baseline in Other PANSS Factors and Subscales at Day 56 and 182
Description: The PANSS provides a total score (sum of the scores of all 30 items) and scores for 3 subscales, the positive subscale (7 items), the negative subscale (7 items), and the general psychopathology subscale (16 items), each rated on a scale of 1 (absent) to 7 (extreme).
Time Frame: Baseline, Day 56 and 182
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER) | Aripiprazole
Number analyzed (Participants) | 112 | 114
Units on a scale
  Baseline: Positive Subscale | 21.5 (4.14) | 22.5 (4.26)
  Change at Day 56: Positive Subscale | -6.4 (4.54) | -6.2 (4.91)
  Change at Day 182: Positive Subscale | -8.0 (5.16) | -8.3 (6.09)
  Baseline: Negative Subscale | 23.8 (4.55) | 24.2 (4.32)
  Change at Day 56: Negative Subscale | -4.2 (4.25) | 4.5 (4.25)
  Change at Day 182: Negative Subscale | -5.7 (5.15) | -6.1 (5.47)
  Baseline: General Psychopathology | 44.3 (7.47) | 45.3 (7.01)
  Change at Day 56: General Psychopathology | -8.7 (7.35) | -9.1 (7.25)
  Change at Day 182: General Psychopathology | -11.9 (9.02) | -12.4 (9.41)

6. Secondary Outcome: Number of Participants With Clinical Stability
Description: Clinical stability is defined as a decrease of 20 percent or more from Baseline in PANSS total score and CGI-S score less than or equal to 4 at Days 56 and 182, no hospitalizations due to psychiatric illness and no emergence of clinically significant suicidal or homicidal ideation during the maintenance phase.
Time Frame: Day 56 and 182
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Paliperidone Extended Release (ER) | Aripiprazole
Number analyzed (Participants) | 112 | 114
Participants | 58 | 68
Statistical Analysis 1: Comparison: Paliperidone Extended Release (ER) vs Aripiprazole; Test type: Superiority or Other; p = 0.296, Cochran-Mantel-Haenszel — Generalized Cochran- Mantel- Haenszel test for row mean score differences controlling for country was used

7. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score at Days 56 and 182
Description: The CGI-S rating scale is a 7-point global assessment that measures the Clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate worsening.
Time Frame: Baseline, Day 56 and 182
Population: as for outcome 2
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER) | Aripiprazole
Number analyzed (Participants) | 112 | 114
Units on a scale
  Baseline | 4.0 [3 to 6] | 4.0 [3 to 6]
  Change at Day 56 | -1.0 [-4 to 0] | -1 [-3 to 1]
  Change at Day 182 | -1.0 [-4 to 1] | -1.0 [-4 to 1]
Statistical Analysis 1: Comparison: Paliperidone Extended Release (ER) vs Aripiprazole; Test type: Superiority or Other; p = 0.843, ANCOVA — Change at Day 56: ANCOVA model on ranks with treatment groups (paliperidone ER, aripiprazole) and country as factors, and baseline value (unranked) as a covariate was used
Statistical Analysis 2: Comparison: Paliperidone Extended Release (ER); Test type: Superiority or Other; p = 0.914, ANCOVA — Change at Day 182: ANCOVA model on ranks with treatment groups (paliperidone ER, aripiprazole) and country as factors, and baseline value (unranked) as a covariate was used

8. Secondary Outcome: Change From Baseline in Personal and Social Performance (PSP) Scores at Day 56 and 182
Description: The PSP scale assesses degree of a participants' dysfunction within 4 domains of behavior: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior. The results of the assessment are converted to a numerical score to rate degree of difficulty (1=absent to 6=very severe) in each of the 4 domains. Based on 4 domains there will be 1 total score (total score ranges from 1 to 100, divided into 10 equal intervals). Participants with score of 71 to 100 have mild degree of difficulty; from 31 to 70, varying degrees of disability; less than or equal to 30, functioning so poorly as to require intensive supervision.
Time Frame: Baseline, Day 56 and Day 182
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Paliperidone Extended Release (ER) | Aripiprazole
Number analyzed (Participants) | 112 | 114
Units on a Scale
  Baseline | 49.8 (10.32) | 49.2 (10.21)
  Change at Day 56 | 12.2 (11.72) | 12.2 (10.17)
  Change at Day 182 | 17.1 (14.46) | 17.1 (14.03)
Statistical Analysis 1: Comparison: Paliperidone Extended Release (ER) vs Aripiprazole; Test type: Superiority or Other; p = 0.895, ANCOVA — Change at Day 56: Analysis of covariance (ANCOVA) model with treatment groups(paliperidone ER, aripiprazole) and country as factors, and baseline value as a covariate was used; LS mean difference = 0.2, 95% CI 2-sided [-2.34 to 2.67], Standard Error of Mean 1.27
Statistical Analysis 2: Comparison: Paliperidone Extended Release (ER) vs Aripiprazole; Test type: Superiority or Other; p = 0.705, ANCOVA — Change at Day 182: Analysis of covariance (ANCOVA) model with treatment groups (paliperidone ER, aripiprazole) and country as factors, and baseline value as a covariate was used; LS mean difference = 0.6, 95% CI 2-sided [-2.64 to 3.89], Standard Error of Mean 1.66

9. Secondary Outcome: Number of Participants With PANSS Response
Description: The PANSS is a 30-item scale with each item rated on a scale of 1 (absent) to 7 (extreme psychopathology), designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Participants with PANSS response were defined as those who achieved greater than or equal to 20 percent or higher reduction from Baseline in the PANSS total score at Day 56 and 182.
Time Frame: Day 56 and 182
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Paliperidone Extended Release (ER) | Aripiprazole
Number analyzed (Participants) | 112 | 114
Participants
  Day 56 | 76 | 87
  Day 182 | 86 | 93
Statistical Analysis 1: Comparison: Paliperidone Extended Release (ER) vs Aripiprazole; Test type: Superiority or Other; p = 0.119, Cochran-Mantel-Haenszel — Day 56: Generalized Cochran-Mantel-Haenszel test for row mean score differences was used
Statistical Analysis 2: Comparison: Paliperidone Extended Release (ER) vs Aripiprazole; Test type: Superiority or Other; p = 0.444, Cochran-Mantel-Haenszel — Day 182: Generalized Cochran-Mantel-Haenszel test for row mean score differences was used

ADVERSE EVENTS:
Time Frame: Baseline up to Week 26
Description: The safety population included all randomly assigned participants who received at least 1 dose of double-blind study drug. A total of 113 participants in the paliperidone ER group and 114 participants in the aripiprazole group received at least 1 dose of double-blind study medication and were included in the safety analysis set.
Arm/Group | Paliperidone Extended Release (ER) | Aripiprazole
Serious Adverse Events (participants affected / at risk) | 7/113 | 7/114
Other Adverse Events (participants affected / at risk) | 63/113 | 50/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Extended Release (ER) (N=113) | Aripiprazole (N=114)
Agitation (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 1 | 4
Schizophrenia, paranoid type (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Extended Release (ER) (N=113) | Aripiprazole (N=114)
Headache (Nervous system disorders) | 12 | 5
Akathisia (Nervous system disorders) | 13 | 9
Somnolence (Nervous system disorders) | 12 | 12
Tremor (Nervous system disorders) | 12 | 11
Sedation (Nervous system disorders) | 6 | 3
Insomnia (Psychiatric disorders) | 6 | 9
Schizophrenia (Psychiatric disorders) | 3 | 10
Vomiting (Gastrointestinal disorders) | 8 | 1
Nausea (Gastrointestinal disorders) | 4 | 7
Weight increased (Investigations) | 12 | 7
Asthenia (General disorders) | 6 | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 7 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator wishes to publish information from the study, a copy of the manuscript must be provided to the Sponsor for review at least 60 days before submission for publication. If requested by the Sponsor, the Investigator will withhold it up to an additional 60 days to allow for filing of a patent application. The Sponsor will not change or suppress the scientific content. For multi-center study, results may not be published before the primary endpoints of a study have been published.